CLINICAL TRIAL: NCT04941131
Title: The Role of Chlorhexidine in Minimizing the Viral Load Among COVID-19 Patients: A Randomized Controlled Clinical Trial
Brief Title: The Role of Chlorhexidine in Minimizing the Viral Load Among COVID-19 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Zuhair Saleh Natto, Head of research unit and associate professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1485
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
Keywords: Mouth Wash; Viral Load
MeSH Terms: conditions — COVID-19 | interventions — chlorhexidine gluconate; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- chlorhexidine digluconate mouthwash (Experimental)
  Interventions: Drug: Chlorhexidine digluconate, povidone iodine
- chlorhexidine digluconate lozenges (Experimental)
  Interventions: Drug: Chlorhexidine digluconate, povidone iodine
- povidone iodine mouthwash (Experimental)
  Interventions: Drug: Chlorhexidine digluconate, povidone iodine
- tap water (No Intervention)

INTERVENTIONS:
Drug: Chlorhexidine digluconate, povidone iodine — This is a mouth wash that can be used over the counter.
  Arms: chlorhexidine digluconate lozenges; chlorhexidine digluconate mouthwash; povidone iodine mouthwash

SUMMARY:
Existing evidence confirmed that saliva and oral cavity to be a reservoir for SARS-CoV-2. In dental clinic aerosol-producing-procedures pose a significant risk for transmission of the infection . It is very important to minimize the risk of transmission in dental office reducing the load of SARS-CoV-2 in saliva if possible, in suspect or conformed cases. Preprocedural mouth rises have been used widely to minimize the number of oral microorganisms. Multiple studies confirmed the efficacy of those mouth rinses in reducing the possibility of transmission of SARS-CoV-2 infection .

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is one of the coronaviruses such as (SARS & MERS) which are commonly known for causing severe respiratory illnesses. SARS-CoV-2 is considered to be the leading cause of coronavirus disease (COVID-19) . On March 11th 2020, the WHO announced that SARS-CoV-2 is a global pandemic. Based on COVID-19 Saudi Arabia Ministry of Health Dashboard, globally, as of April 5th 2021, there have been more than 131 million confirmed cases of the disease including more than 2 million deaths. Nationally, as of April 5th 2021, there have been 392,682 confirmed cases including 6,697 deaths .

The diagnosis of COVID-19 involves molecular testing which is the gold standard and the WHO most recommended method of diagnosis. SARS-CoV-2 seemed to be very contagious and the chances of its transmission even before any symptoms occur are very high. It has been documented that COVID-19 disease incubation period to range between 1-14 days, most reported to be between 3 to 7 days with some evidence suggested the incubation period of 5 days. Evidence concerned about the spread of infection due to missed screened cases especially when individuals are unaware of their infection status and didn't show any symptoms yet.

Existing evidence confirmed that saliva and oral cavity to be a reservoir for SARS-CoV-2 . Multiple studies suggested SARS-CoV-2 to be airborne infection, and get transmitted through aerosols. In dental clinic aerosol-producing-procedures pose a significant risk for transmission of the infection. It is very important to minimize the risk of transmission in dental office reducing the load of SARS-CoV-2 in saliva if possible, in suspect or conformed cases. Preprocedural mouth rises have been used widely to minimize the number of oral microorganisms. Multiple studies confirmed the efficacy of those mouth rinses in reducing the possibility of transmission of SARS-CoV-2 infection .

The aim of our study is to determine the efficacy of different mouthwash in reducing the SARS-CoV-2 viral load in saliva of COVID-19 confirmed cases compared with tap water.

The objectives of the study are to determine the viral load, assess the cases clinical information & disease manifestation, plus the cases demographic characteristics believed to have an influence on the disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

* A history of positive nasal swabs for SARS-CoV-2 based on reverse-transcription polymerase chain reaction (RT-PCR) assays.

Exclusion Criteria:

* History of allergy to any of the products that will be used
* known pregnancy
* Renal failure

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University , Faculty of Dentistry, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Natto ZS, Bakhrebah MA, Afeef M, Al-Harbi S, Nassar MS, Alhetheel AF, Ashi H. The short-term effect of different chlorhexidine forms versus povidone iodine mouth rinse in minimizing the oral SARS-CoV-2 viral load: An open label randomized controlled clinical trial study. Medicine (Baltimore). 2022 Jul 29;101(30):e28925. doi: 10.1097/MD.0000000000028925. PMID 35905275

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorhexidine Digluconate Mouthwash; Chlorhexidine Digluconate Lozenges; Povidone Iodine Mouthwash: This is a mouth wash that can be used over the counter.
- Tap Water: It is regular tap water
Period: Overall Study
Arm/Group | Chlorhexidine Digluconate Mouthwash | Chlorhexidine Digluconate Lozenges | Povidone Iodine Mouthwash | Tap Water
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Digluconate Mouthwash | Chlorhexidine Digluconate Lozenges | Povidone Iodine Mouthwash | Tap Water | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: Year] — Population: We have 15 participants per group assigned in the protocol. The range was between 12 to 15 max. We were able to get the max in each group
  Year | 37.80 (11.24) | 36.20 (13.21) | 33.86 (10.29) | 41.73 (17.14) | 37.40 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We have 15 participants per group assigned in the protocol. The range was between 12 to 15 max. We were able to get the max in each group
  Participants
    Female | 7 | 3 | 4 | 4 | 18
    Male | 8 | 12 | 11 | 11 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
E genes [Mean (Standard Deviation); unit: Cycle] — Population: We have 15 participants per group assigned in the protocol. The range was between 12 to 15 max. We were able to get the max in each group
  Cycle | 26.23 (7.37) | 26.14 (5.98) | 25.85 (6.33) | 27.59 (5.01) | 26.44 (6.01)
S genes [Mean (Standard Deviation); unit: Cycle] — Population: We have 15 participants per group assigned in the protocol. The range was between 12 to 15 max. We were able to get the max in each group
  Cycle | 25.03 (6.63) | 24.83 (5.13) | 25.18 (6.35) | 26.11 (4.04) | 25.24 (5.53)

OUTCOME MEASURES:

1. Primary Outcome: E Genes
Description: Gene viral load serves as a proxy measure for the presence and quantity of SARS-CoV-2 virus in patient samples. Since the E gene is expressed early and reliably during viral replication, changes in its detected levels reflect the dynamics of viral presence. Quantified using RT-qPCR, with results expressed as cycle threshold (Ct) values-the number of amplification cycles required to detect the gene above background levels. Lower Ct values indicate higher viral loads.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Cycle
Arm/Group | Chlorhexidine Digluconate Mouthwash | Chlorhexidine Digluconate Lozenges | Povidone Iodine Mouthwash | Tap Water
Number analyzed (Participants) | 15 | 15 | 15 | 15
Cycle | 28.50 (5.21) | 27.33 (4.9) | 30.28 (6.33) | 27.80 (4.33)

2. Secondary Outcome: S Genes
Description: Gene viral load serves as a proxy measure for the presence and quantity of SARS-CoV-2 virus in patient samples. Since the S gene is expressed early and reliably during viral replication, changes in its detected levels reflect the dynamics of viral presence. Quantified using RT-qPCR, with results expressed as cycle threshold (Ct) values-the number of amplification cycles required to detect the gene above background levels. Lower Ct values indicate higher viral loads.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Cycle
Arm/Group | Chlorhexidine Digluconate Mouthwash | Chlorhexidine Digluconate Lozenges | Povidone Iodine Mouthwash | Tap Water
Number analyzed (Participants) | 15 | 15 | 15 | 15
Cycle | 27.86 (5.89) | 26.74 (5.27) | 28.09 (6.37) | 27.87 (3.83)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Tap Water: Regular water
Arm/Group | Chlorhexidine Digluconate Mouthwash | Chlorhexidine Digluconate Lozenges | Povidone Iodine Mouthwash | Tap Water
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT04941131/Prot_SAP_002.pdf